CLINICAL TRIAL: NCT03109327
Title: Investigating the Clinical Utility of the MDS Test for the Oncogenic Activity in Nevi Suspected of Being Melanoma
Brief Title: Investigating the Clinical Utility of the MDS
Acronym: OMS002_UK
Status: Completed | Type: Observational
Sponsor: Orlucent, Inc (Industry)
Collaborators: NHS Lanarkshire (Other Government); NHS Tayside (Other Government); NHS Greater Glasgow and Clyde (Other); University Hospitals, Leicester (Other); University of Dundee (Other)
Responsible Party: Sponsor
Other Study IDs: OMS002_UK
Record Dates: First submitted 2017-03-08; First posted 2017-04-12 (Actual); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Skin Lesion; Melanoma; Moles
MeSH Terms: conditions — Melanoma; Nevus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Urgent Excision: Subjects with moles suspicious of melanoma and are scheduled for an urgent excision.
  Interventions: Diagnostic Test: Melanoma Detection System -MDS
- Non-urgent Excision: Subjects with moles not-suspicious of melanoma and are scheduled for a non urgent excision.
  Interventions: Diagnostic Test: Melanoma Detection System -MDS

INTERVENTIONS:
Diagnostic Test: Melanoma Detection System -MDS — Imaging of lesion using the MDS test.
  Other Names: MDS

SUMMARY:
The purpose of this study is to establish the clinical utility of the Melanoma Detection System (MDS).

DETAILED DESCRIPTION:
The purpose of this study is to establish the clinical utility of the MDS while continuing to evaluate the safety and performance of the MDS in patients with skin lesions who are referred to secondary care clinics for evaluation, whose lesions (moles) are suspicious for melanoma.

ELIGIBILITY:
Inclusion Criteria:

1. Lesion has one or more of the ABCDE features and is recommended for excision.
2. Lesion has at least 1 cm of skin around it that is accessible to the MDS.
3. Patient is at least 18 years old.
4. Patient is capable of giving written informed consent.
5. Lesion is scheduled for primary excision.

Exclusion Criteria:

1. Lesion is less than one centimetre from the eyes.
2. Lesion is on the palms of the hands or soles of the feet.
3. Lesion is mucosal.
4. Lesion is ulcerated.
5. Patient is pregnant.
6. Low patient study procedure compliance.
7. Patient who is mentally or physically unable to comply with all aspects of the study.
8. Patient is undergoing chemotherapy.
9. Patient has known sensitivity to fluorescent dyes.
10. Ink marking on or adjacent to lesion.
11. Lesions larger than 20mm or too large to allow imaging.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects referred to a specialist for possible presence of melanoma in skin lesions.
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Utility of the MDS in determining urgent or non-urgent excision of moles. | 1 day
  The MDS will provide a score that reflects the possibility for the presence of melanoma in moles. The score will be used together with clinical evaluation.

SECONDARY OUTCOMES:
Does the MDS have an additive value to clinical evaluation of moles. | 1 day
  Does the MDS system provide superior results when compared to clinical evaluation.

OTHER OUTCOMES:
User feedback for clinical use of the MDS in the clinical management of moles. | 1 day
  To gain feedback from users on how to best incorporate the MDS testing procedure in the clinical setting.

CONTACTS AND LOCATIONS:
Locations (1):
- NHS Lanarkshire, Monklands Hospital, Airdrie, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided